CLINICAL TRIAL: NCT03151421
Title: Measuring for Change: Air Quality Feedback to Reduce Second-hand Smoke (SHS) Exposure in the Home
Brief Title: Air Quality Feedback to Reduce Second-hand Smoke (SHS) Exposure in the Home
Acronym: TackSHSWP4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: University of Aberdeen (Other); Istituto per lo Studio, la Prevenzione e la Rete Oncologica (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Hellenic Cancer Society (Other); Public Health Agency of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TackSHS WP4
Record Dates: First submitted 2017-03-30; First posted 2017-05-12 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Second Hand Tobacco Smoke; Tobacco Smoking; Tobacco Use
Keywords: air quality feedback; second-hand smoke; passive smoking; exposure to second-hand smoke; second-hand smoke exposure prevention
MeSH Terms: conditions — Tobacco Smoking; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home air quality monitoring and feedback (Experimental): Home air quality monitoring and feedback
  Interventions: Behavioral: Home air quality monitoring and feedback

INTERVENTIONS:
Behavioral: Home air quality monitoring and feedback — Two-hundred smokers (50 in each country) will be recruited and offered low-cost, simple to operate particle counting instruments to measure and log SHS levels in their home for a period of 30 days. During this time near real-time, personalised feedback will be provided to, and discussed with, the smoker along with target-setting and exploration of suitable methods of behaviour-change. Feedback will be given via text message to mobile phones, emails and personal voicecalls. A final visit will gather data on changes made while a proportion of participants (10-20%) in each country will take part in a further qualitative interview by phone to gather data on their experience of the intervention.

SUMMARY:
This is a European study which is part of a larger research project (The TackSHS project) funded by the European Union's Horizon 2020 Research and Innovation Programme (Grant Agreement No 681040) and led by the Catalan Institute of Oncology.

This study will examine the efficacy of using personalised air quality measurements in homes of smokers to encourage behaviour-change towards having a smoke-free home environment. Building on recent quantitative and qualitative work showing that feedback of second-hand smoke (SHS) measurement information can help motivate smokers to change their behaviour. This study will develop a targeted intervention for use with socio-economically deprived smokers in four countries (Scotland, Spain, Greece, Italy) across the EU. Two-hundred smokers (50 in each country) will be recruited and offered low-cost, simple to operate particle counting instruments to measure and log SHS levels in their home for a period of 30 days. During this time near real-time, personalised feedback will be provided to, and discussed with, the smoker along with target-setting and exploration of suitable methods of behaviour-change. Feedback will be given via text message to mobile phones, emails and personal voice calls. A final visit will gather data on changes made while a proportion of participants (10-20%) in each country will take part in a further qualitative interview by phone to gather data on their experience of the intervention.

Study outcomes will include quantitative measures such as changes in average and maximum fine particulate matter (PM2.5) concentrations and self-declared household smoking rules, while qualitative data will be gathered using questionnaire and interview to explore what elements of the intervention were useful/unhelpful, particularly well/poorly understood, and what were the barriers for those who did not make changes. This WP will provide a comprehensive database of baseline measurements of SHS concentrations in home settings from across the EU with the potential to generate over 8 million minutes of measurements of household air quality. Analysis of the differences by country and possible determinants of exposure will be carried out.

DETAILED DESCRIPTION:
Main Aim:

To create a smoke-free environment for children of parents who smoke, by having parents exchange ineffective strategies to create a smoke-free environment (e.g. smoking in another room in the house) for effective strategies (e.g. smoking outside, delaying smoking, quitting smoking).

Sub Aim:

To test the feasibility and effectiveness of using new, internet-connected air quality monitors to record and upload air quality information as part of an educational intervention on the effects of smoking on household air quality.

Research Questions:

1. Can low-cost, internet-connected air quality monitors effectively detect second-hand smoke-related PM2.5 and relay this information to researchers?
2. Can delivering this information together with advice about keeping homes smoke-free on a daily basis over a month promote behaviour change?
3. Is providing remote feedback on air quality levels a feasible method of engaging with parents living in areas of socio-economic deprivation?

STUDY DESIGN

This is a multi-country study using a single arm pre-test/post-test design.

STUDY SETTINGS

The study will be carried out in smokers' homes in areas of multiple deprivation in Greece, Italy, Spain and the United Kingdom. These countries have variable rates of smoking prevalence and a range of smoke-free places legislation, smoke-free homes policies and therefore varying prevalence of childhood exposure to second-hand smoke.

RECRUITMENT

Participants will be recruited using targeted adverts and leaflets within public sector and third sector environments in socio-economically deprived areas. Environments used to recruit may include nurseries, libraries, family centres and other family directed help services within the community. Where necessary direct advertising using traditional or social media may also be employed. Participants will be able to express interest in taking part in the study by contacting the research team by phone, email or text.

When a contact is made the research team will then initiate a brief telephone conversation to address any queries and determine eligibility for inclusion in the study.

Once the potential participant is identified as suitable for inclusion and verbal consent has been given then a Participant Information Sheet (PIS) will be sent to the participant by email. Participants will have a minimum of 48 hours to consider the information they have been sent, after which one of the researchers will contact them again to check whether they are still happy to take part in the study, and if so, to arrange a suitable time for the first home visit to install the Air Quality Monitor (AQM) to take place.

Participants will be given a £10 (or equivalent in Euros) shopping voucher for taking take part in the study, and a further £10 if they decide to take part in the qualitative interview. These vouchers acknowledge any minimal electricity/WiFi costs incurred as a result of taking part in the study, and provide a means of thanking participants' for their time in participating.

HOUSEHOLD VISITS

Informed, signed consent will be obtained at the beginning of the visit based on the previously obtained PIS.

The AQM will be installed in the main living area of the home by the visiting researcher. The monitor will be placed in a position that should be elevated at between 0.5-1.5m from the floor, and at least 0.5m from a wall, window or door. The AQM will require a functioning electrical outlet.

The AQM will be tethered to the household WiFi network. If the participant does not have wireless broadband in their home, a pre-paid 3g/4g WiFi router will be assigned and installed. Where a pre-paid 3g/4g WiFi router is installed this will not permit any other devices to use the connection and will solely be for transfer of data from the AQM.

"Knowledge, Beliefs & Attitudes" module previously developed for the AFRESH programme (http://www.smokefreehomes.network/) will be explored with the smoker and the baseline questionnaire completed. This whole process should take approximately 45 minutes.

The AQM will then be left in situ for 30 days.

DATA SOURCES

Air quality monitoring Fine particulate matter will be monitored in each participant's home.

The Foobot (www.foobot.io) AQM will be used in this intervention. The Foobot is a low-cost monitor containing particulate matter (PM), volatile organic compound (VOC), temperature and humidity sensors. For the purposes of this study, the PM sensor will be used, as fine PM (PM2.5) is an effective marker for the presence of SHS. Data such as VOC, temperature and humidity may be utilised to help develop a predictive algorithm to help with the differentiation of SHS from other sources of fine PM.

The Foobot's PM sensor has been tested internally in lab trials with second-hand smoke and other air pollutants. Each participating institute will be assigned 8 Foobot instruments providing them with the maximal capability of measuring in 8 homes per month.

Questionnaires

Each participant will be asked to complete a baseline questionnaire at the first visit from the researcher. This questionnaire will ask about their home's inhabitants, their smoking behaviours, smoking rules for others in the home and questions and their intention to change smoking behaviours in the home. This will validate their inclusion in the study.

A follow-up questionnaire will gather data on changes in smoking rules in the home and views on the intervention as an outcome measure. This questionnaire will be delivered at the end of the 30 day intervention period.

Qualitative interviews

Between 4 and 8 participants in each country will be recruited to take part in semi-structured interviews to discuss their experience of the intervention. A shopping voucher of value £10 will be provided to reimburse participants for their time. The consent form and interview topic guide for this work were adopted from AFRESH Programme (see above).

DATA MANAGEMENT

Data will be stored on Foobot company servers and downloaded each day using a custom programme developed by University of Aberdeen researchers No identifying information on the participants will be stored on the Foobot company servers, but researchers will have access to personal information, including name, address, telephone number and email address.

Email and text message feedback will be sent using the custom developed programme or (where appropriate or required) personal accounts. The Clockwork SMS API (www.clockworksms.com) will be used to send SMS messages over the internet, while university or insitutional email accounts will be used to send emails.

Personal information will be treated as confidential in line with relevant country and EU data protection legislation. Consent forms and questionnaires, once collected, will be posted (by secure mail) to the University of Aberdeen and retained in a locked filing cabinet for seven years.

PERSONALISED FEEDBACK

At the end of the baseline measurement week the research team will initiate a series of contacts with the participant for the following 3 weeks.

Firstly a feedback text will be sent to the participant's mobile phone providing them with details of their average levels of PM in the previous week (day 8). An email with a link to their detailed weekly graph will also be provided on this day. This will be followed up the next day (day 9) with a telephone call at a pre-arranged time to discuss their results and to talk through facilitators, barriers and solutions, and planning around 'What if…' scenarios.

From day 9 onwards daily text message results with supportive comments and suggestions will be sent to the participant's mobile phone (days 9-29). Support phone calls providing more detailed feedback and revisiting AFRESH modules "Barriers, solutions and facilitators to creating a smoke-free home" and "Planning for creating a smoke-free home" will be given after week 2 (day 16) and 3 (day 23). Weekly graphs/reports will be sent by email to the participant the day prior to these telephone conversations (day 15 and 22).

On day 30 the researcher will visit with personalised feedback covering the whole one-month period grouped in to the 4 previous weekly blocks. Discussion will be around progress achieved and plans for the future.

LOCAL VARIATION

This study will be carried out in Scotland (the UK), Catalonia (Spain), Greece, and Italy. The general protocol will be similar in all four countries with some minor changes to the recruitment process depending on local and cultural norms. Consent forms, questionnaires, the PIS and email and text messages will be translated into local languages as required.

POWER CALCULATION

At an individual country level the study will recruit 50 households to participate. Using PM2.5 concentrations in the final 7 days of the 30 day measurement period as the study primary outcome measure, and assuming that participants achieve a 50% reduction in fine particle levels compared to the baseline measurements in days 1-7, a sample of 35 will give a power of >80% with an alpha level of 0.05. This is based on data gathered from the First Steps to Smoke-Free (FS2SE) project where it wasfound an average baseline PM2.5 concentration of 67.5 µg/m3 (SD 79.7 µg/m3). Recruiting 50 subjects will thus provide sufficient numbers assuming drop-out is <12% (broadly in line with investigators' experience in the FS2SF study where 15 participants were lost from the 117 that completed baseline). A 50% reduction in the mean PM2.5 value is realistic in terms of the size of change seen in other study, REFRESH, (geometric mean fell from 19 to 11 µg/m3 at one-month). Pooled across the 4 study sites (assuming similar exposures) a total study size of 175 homes completing the 30 day study would provide 80% power to detect a decrease of 22% in PM2.5 concentrations.

STATISTICAL ANALYSIS

Arithmetic mean concentrations of PM2.5 will be calculated for homes over the days 1-7, days 23-29 and whole sampling time, and presented with standard deviations and ranges. All-sample mean and median concentrations over each time period will be calculated and compared for each country.

A first descriptive analysis will be conducted for all outcomes included in the study. Categorical variables will be described by raw frequencies and percentages and continuous variables will be described by means and standard deviations or medians and interquartile range (IQR).

Medians and IQR of PM2.5 concentrations will be calculated by country and overall for the complete intervention group. Box-plots will be used to visualize the distribution of PM2.5 concentrations. A separate secondary analysis of data by country will also be conducted.

Analysis will be conducted using Microsoft Excel 2013 and IBM SPSS v24.

ETHICS

This study will be conducted in line with the Good Clinical Practice guidelines of the Declaration of Helsinki, along with applicable EU and local legislation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18 years or over) who smokes inside their home on a daily basis
2. Takes care of a child (16 years old or under) in their home at least once per week
3. Lives in a SIMD quintile 1 or 2 postcode or equivalent (i.e. within 40% most deprived households in their country)
4. Does not plan to move home in the next 2 months
5. Is at the contemplative stage regarding having a smoke-free home and indicates that they feel it would be possible for their home to go smoke-free
6. Has a personal mobile phone, email address and some form of regular access to the internet (either by computer or smartphone)

Exclusion Criteria:

1. Persons with low literacy level that would prevent understanding and following study instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in air quality (pre-/post-intervention) | The intervention will last 1 month. Comparison of differences in PM2.5 average concentrations during the first week of intervention (day 1-7) and the last one (day 23-29)
  Arithmetic mean concentrations of PM2.5 will be calculated for homes over the days 1-7, days 23-29 and whole sampling time, and presented with standard deviations and ranges.

SECONDARY OUTCOMES:
Changes in self-declared household smoking rules (pre-/post-intervention) | Pre-/post intervention (30 days)
  Each participant will be asked to complete a baseline questionnaire at the first visit from the researcher. This questionnaire will ask about their home's inhabitants, their smoking behaviours, smoking rules for others in the home and their intention to change smoking behaviours in the home. A follow-up questionnaire will gather data on changes in smoking rules in the home. This questionnaire will be delivered at the end of the 30 day intervention period.
Effectiveness of the intervention (self-declared) | After the 30 days of the intervention (one time-point measurement)
  Between 4 and 8 participants in each country will be recruited to take part in semi-structured interviews to discuss their experience of the intervention. Qualitative data will be gathered to explore what elements of the intervention were useful/unhelpful, particularly well/poorly understood, and what were the barriers for those who did not make changes.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Semple, PhD, Principal Investigator — University of Aberdeen, Respiratory Group, Division of Applied Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: TackSHS Project at CORDIS — https://cordis.europa.eu/project/rcn/198790/factsheet/en